CLINICAL TRIAL: NCT01296633
Title: Medtable: An Electronic Medical Record (EMR) Strategy to Promote Patient Medication Understanding and Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Northwestern University (Other); OSF Healthcare System (Other)
Responsible Party: Principal Investigator, Dan Morrow, PhD, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01NR011300-01A1 (NIH)
Record Dates: First submitted 2011-01-06; First posted 2011-02-15 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus
Keywords: health literacy; patient education; medication adherence; patient/provider communication; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medtable (Experimental): The Medtable is a patient education tool used for collaborative planning. The Medtable focuses patients on how to take their medication and prompts them to anchor this task to familiar routines. The tool serves as an external workspace that helps provider and patient jointly visualize how to integrate constraints from medications (e.g., which can be taken together; dose spacing) and patients' routine (e.g., typical meal times) in order to create an optimal daily schedule. The completed Medtable shows providers how patients are thinking about taking their medications, allowing them to clear up any confusion. It encourages teach-back and teach-to-goal strategies recommended for patients with low health literacy. Completing the Medtable helps patients implement as well as create plans by encouraging them to think about when and where they will actually take their medication. It also provides a template developed with their providers that could help patients load pill organizers at home.
  Interventions: Behavioral: Medtable
- Usual care (Active Comparator): Patients in the usual care condition at both research sites will receive the medication counseling and communication that is standard of care at these sites. This includes a medication reconciliation process, where patients are given a card with list of medications that is periodically checked. This provides an opportunity for providers to correct patient knowledge of their medications, and is similar to the process of creating a list for the Medtable. However, the Medtable also encourages patients and providers to collaborate in order to organize this list in terms of the patient's routine to create a patient-specific, concrete plan for taking the medications.
  Interventions: Behavioral: Medtable

INTERVENTIONS:
Behavioral: Medtable — Nurse works with patient to reconcile EMR-based medication list and load list into Medtable. Nurse uses Medtable with patient to develop plans for taking medications. Patient completes Medtable columns to identify when routine activities are performed during the day. Nurse discusses medications with patient: what the medication is called, used for, etc. Nurse and patient jointly develop the schedule by choosing times to take each medication. These times are entered into corresponding cells of the Medtable. Nurse corrects any mistakes (e.g., times that would conflict with dose spacing requirements). Nurse asks patient to review to ensure patient understands key facts and that drug interactions or other restrictions are addressed, using collaborative inquiry, teach-back, and teach-to-goal strategies. Patient takes home a hardcopy of the Medtable schedule to guide adherence. An updated e-copy is integrated with patient's record in the EMR.

SUMMARY:
The broad goal of this project is to improve knowledge of and adherence to medication regimens and health outcomes among adults with type 2 diabetes or other metabolic disorders. These patients have complex self-care needs, but limited literacy and cognitive skills to meet these needs. Medication error is widespread and costly, and often associated with inadequate patient knowledge about medication, especially among chronically ill adults with limited health literacy. Inadequate knowledge is often traced to limited communication with providers, in part because of barriers such as limited patient contact time and communication training, and lack of system-level support for consistent use of patient-centered strategies. There is a need to leverage information technology (IT) to provide system-based support for patient-centered communication. The investigators will evaluate an Electronic Medical Record (EMR)-based tool (the Medtable) to support provider/patient communication and improve medication knowledge, adherence, and health outcomes among chronically ill adults with complex medication regimens. A paper-based Medtable has been found to help older adults create accurate medication schedules in a simulated patient/provider communication task (Morrow et al., 2008). Benefits for patients should be enhanced if the Medtable is integrated with an EMR, giving providers ready access to relevant background information and current medication lists that patients can update, so providers can generate and tailor the Medtable for a diverse set of patients. This system provides an integrated approach to patient education about medications, from prescribing to counseling during office visits. As a result, patients would not only understand how to take their medications, but develop concrete plans for doing so. Specific aims of the project are: 1) Refine the Medtable prototype for use in an EMR environment. This includes developing protocols for generating patient-specific Medtables and educating providers to use them in medical encounters. 2) Evaluate the Medtable's impact on patient care processes and outcomes. The investigators will test the following hypothesis about communication processes: H1) Patients in the intervention condition will be more satisfied with communication about medication than patients in the usual care condition. The investigators will also test the following hypotheses about patient outcomes: Compared to usual care patients, patients receiving the Medtable intervention will: H2) know more about their medications; H3) adhere more accurately to their medication regimens; H4) more likely have blood glucose (glycosylated hemoglobin, HbA1c) levels in the target range. Aim 1 will be accomplished by interviewing physicians and their patients as the system is refined to ensure ease of using the system, and by collecting preliminary evidence that the Medtable improves patient/provider communication. After establishing initial feasibility and ensuring provider acceptance of the system, Aim 2 is addressed by a randomized trial at the general internal medicine clinics in Chicago and Peoria (IL), comparing patients who use the Medtable with their providers to those receiving usual care.

DETAILED DESCRIPTION:
The investigators will integrate the paper-based Medtable into the electronic medical record (EMR) system at the two research sites and evaluate whether this EMR-based tool improves patient/provider communication, patients' medication knowledge, and health outcomes. The EMR will produce Medtables that summarize patients' complex medication schedules with simple, direct language. The Medtable will be used interactively by providers and patients with complex self-care needs in order to create patient-specific adherence plans. Thus, the EMR-based Medtable will help integrate patient-centered communication practices into the prescribing and counseling phases of the medication use process. The Medtable will be used by nurses as part of medication reconciliation and counseling at general internal medicine clinics in Chicago and Peoria that provide routine care to outpatients with complex health care needs. The researchers seek to investigate adults who take complex medication regimens to treat their chronic illness and struggle with self-care (patients with diabetes or other metabolic disorders who have glycosylated hemoglobin (HbA1c) levels higher than 7.0). Patients varying in age, education, and literacy/cognitive abilities will be recruited in order to explore whether the Medtable especially benefits those with lower health literacy, reducing literacy-related differences in medication knowledge, adherence, and outcomes.

In Phase I, the investigators develop the EMR-based Medtable (Year 1). To collect initial feasibility data, the Medtable will be integrated into the EMR-supported practice of several physicians at general internal medicine clinics serving diverse patient populations at Northwestern Medical Foundation (Chicago) and OSF Medical Group (Peoria). Both sites use the Epic EMR system (Epic Systems Corp, Verona, WI). Through interviews and questionnaires the researchers will assess ease of using the Medtable as part of routine clinical practice. Preliminary data about physician adoption (e.g., frequency of generating Medtables for patients) will be collected. Patients of these physicians will be interviewed about ease of using the Medtable and whether it improves satisfaction with patient/provider communication, knowledge, and ability to take their medications. Medtable interface and protocol will be iteratively refined in response to provider and patient feedback.

In Phase II, the researchers will use a randomized trial to evaluate the efficacy of the EMR-based Medtable as a provider/patient collaboration tool for improving patient knowledge and outcomes (Years 2-3).

The researchers will use a random process to assign patients at each clinic site to the Medtable intervention or to usual care condition. For the intervention, the Medtable will be integrated into routine patient activities during office visits: a) during intake, intervention nurses generate the Medtable via the EMR and reconcile medication lists by working with patients; b) at the end of the visit, the nurses and patients use the Medtable to develop easy to understand and implement patient-specific plans for taking the medications. Patients take home a hardcopy of their Medtable-based schedule to guide adherence, and the electronic copy is integrated with the patient EMR.

Outcome measures (for both intervention and usual care patients) are medication knowledge (immediately, 3, and 6 months after the Medtable intervention is introduced), adherence (baseline, 3 and 6 months), and HbA1c level (baseline, 3, 6, 9 and 12 months). Finally, data about how the Medtable is used will be collected, including frequency of generating the Medtable during patient visits, and time required to generate and use the Medtable during routine office visits.

ELIGIBILITY:
Providers:

Physicians will be eligible if they have a significant proportion of patients age 40 or older with metabolic disorders.

Inclusion criteria for nurses will be:

* a current RN, LPN certificate or BSN degree
* practicing at least 10 hours weekly
* providing primary care to adults over age 40 years with chronic illness

This should ensure that we recruit physicians and nurses who teach patients about medication as part of their routine responsibilities.

Patient Participants:

Community-dwelling adults who are patients of participating providers and who meet the following inclusion criteria will participate:

* age 40 and older
* native speaker of English or English speaker before age of 6
* no physical or cognitive impairments that could limit participation (e.g., stroke in the last 3 years, current cancer treatment involving radiation or chemotherapy)
* score of 24 or higher on the Mini Mental State Exam (Folstein, Folstein, & McHugh, 1975)
* no severe visual impairment (<20/50 corrected vision) or auditory impairment that would limit participation
* diagnosis of type 2 diabetes or other metabolic disorders (they are also likely to have other chronic illnesses such as hypertension)
* taking at least 5 prescribed medications
* HbA1c level of 7.0 or higher

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 674 (Actual)
Dates: Start 2011-02; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Medication regimen knowledge | One year

SECONDARY OUTCOMES:
Medication adherence | One year
Patient satisfaction with information about medications | One year
Glycosylated hemoglobin blood test (HBA1c) | One year
Patient-provider communication assessment | One day

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G Morrow, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (2):
- United States (2):
  - Northwestern Medical Faculty Foundation Clinic of Northwestern University, Chicago, Illinois
  - OSF Medical Group of OSF Saint Francis Medical Center, Peoria, Illinois

REFERENCES:
- [Background] Health literacy: report of the Council on Scientific Affairs. Ad Hoc Committee on Health Literacy for the Council on Scientific Affairs, American Medical Association. JAMA. 1999 Feb 10;281(6):552-7. PMID 10022112
- [Background] Altman DE, Clancy C, Blendon RJ. Improving patient safety--five years after the IOM report. N Engl J Med. 2004 Nov 11;351(20):2041-3. doi: 10.1056/NEJMp048243. No abstract available. PMID 15537902
- [Background] American Diabetes Association. Standards of medical care in diabetes--2009. Diabetes Care. 2009 Jan;32 Suppl 1(Suppl 1):S13-61. doi: 10.2337/dc09-S013. No abstract available. PMID 19118286
- [Background] Baker DW, Gazmararian JA, Sudano J, Patterson M. The association between age and health literacy among elderly persons. J Gerontol B Psychol Sci Soc Sci. 2000 Nov;55(6):S368-74. doi: 10.1093/geronb/55.6.s368. PMID 11078114
- [Background] Baker DW, Wolf MS, Feinglass J, Thompson JA, Gazmararian JA, Huang J. Health literacy and mortality among elderly persons. Arch Intern Med. 2007 Jul 23;167(14):1503-9. doi: 10.1001/archinte.167.14.1503. PMID 17646604
- [Background] Baker DW, Wolf MS, Feinglass J, Thompson JA. Health literacy, cognitive abilities, and mortality among elderly persons. J Gen Intern Med. 2008 Jun;23(6):723-6. doi: 10.1007/s11606-008-0566-4. Epub 2008 Mar 11. PMID 18330654
- [Background] Castro CM, Wilson C, Wang F, Schillinger D. Babel babble: physicians' use of unclarified medical jargon with patients. Am J Health Behav. 2007 Sep-Oct;31 Suppl 1:S85-95. doi: 10.5555/ajhb.2007.31.supp.S85. PMID 17931142
- [Background] Davis TC, Wolf MS, Bass PF 3rd, Middlebrooks M, Kennen E, Baker DW, Bennett CL, Durazo-Arvizu R, Bocchini A, Savory S, Parker RM. Low literacy impairs comprehension of prescription drug warning labels. J Gen Intern Med. 2006 Aug;21(8):847-51. doi: 10.1111/j.1525-1497.2006.00529.x. PMID 16881945
- [Background] Davis TC, Wolf MS, Bass PF 3rd, Thompson JA, Tilson HH, Neuberger M, Parker RM. Literacy and misunderstanding prescription drug labels. Ann Intern Med. 2006 Dec 19;145(12):887-94. doi: 10.7326/0003-4819-145-12-200612190-00144. Epub 2006 Nov 29. PMID 17135578
- [Background] Dewalt DA, Berkman ND, Sheridan S, Lohr KN, Pignone MP. Literacy and health outcomes: a systematic review of the literature. J Gen Intern Med. 2004 Dec;19(12):1228-39. doi: 10.1111/j.1525-1497.2004.40153.x. PMID 15610334
- [Background] DeWalt DA, Malone RM, Bryant ME, Kosnar MC, Corr KE, Rothman RL, Sueta CA, Pignone MP. A heart failure self-management program for patients of all literacy levels: a randomized, controlled trial [ISRCTN11535170]. BMC Health Serv Res. 2006 Mar 13;6:30. doi: 10.1186/1472-6963-6-30. PMID 16533388
- [Background] Forster AJ, Murff HJ, Peterson JF, Gandhi TK, Bates DW. The incidence and severity of adverse events affecting patients after discharge from the hospital. Ann Intern Med. 2003 Feb 4;138(3):161-7. doi: 10.7326/0003-4819-138-3-200302040-00007. PMID 12558354
- [Background] Gazmararian JA, Baker DW, Williams MV, Parker RM, Scott TL, Green DC, Fehrenbach SN, Ren J, Koplan JP. Health literacy among Medicare enrollees in a managed care organization. JAMA. 1999 Feb 10;281(6):545-51. doi: 10.1001/jama.281.6.545. PMID 10022111
- [Background] Houts PS, Doak CC, Doak LG, Loscalzo MJ. The role of pictures in improving health communication: a review of research on attention, comprehension, recall, and adherence. Patient Educ Couns. 2006 May;61(2):173-90. doi: 10.1016/j.pec.2005.05.004. Epub 2005 Aug 24. PMID 16122896
- [Background] Kripalani S, Robertson R, Love-Ghaffari MH, Henderson LE, Praska J, Strawder A, Katz MG, Jacobson TA. Development of an illustrated medication schedule as a low-literacy patient education tool. Patient Educ Couns. 2007 Jun;66(3):368-77. doi: 10.1016/j.pec.2007.01.020. Epub 2007 Mar 6. PMID 17344015
- [Background] Levinthal BR, Morrow DG, Tu W, Wu J, Murray MD. Cognition and health literacy in patients with hypertension. J Gen Intern Med. 2008 Aug;23(8):1172-6. doi: 10.1007/s11606-008-0612-2. Epub 2008 May 6. PMID 18459011
- [Background] Makoul G. Essential elements of communication in medical encounters: the Kalamazoo consensus statement. Acad Med. 2001 Apr;76(4):390-3. doi: 10.1097/00001888-200104000-00021. PMID 11299158
- [Background] Morrow D. Improving consultations between health-care professionals and older clients: implications for pharmacists. Int J Aging Hum Dev. 1997;44(1):47-72. doi: 10.2190/GQX9-F4UJ-5RQ2-N1YD. PMID 9131381
- [Background] Morrow D, Carver LM, Leirer VO, Tanke ED. Medication schemas and memory for automated telephone messages. Hum Factors. 2000 Winter;42(4):523-40. doi: 10.1518/001872000779698042. PMID 11324848
- [Background] Morrow D, Clark D, Tu W, Wu J, Weiner M, Steinley D, Murray MD. Correlates of health literacy in patients with chronic heart failure. Gerontologist. 2006 Oct;46(5):669-76. doi: 10.1093/geront/46.5.669. PMID 17050758
- [Background] Morrow DG, Hier CM, Menard WE, Leirer VO. Icons improve older and younger adults' comprehension of medication information. J Gerontol B Psychol Sci Soc Sci. 1998 Jul;53(4):P240-54. doi: 10.1093/geronb/53b.4.p240. PMID 9679516
- [Background] Morrow DG, Leirer VO, Andrassy JM, Hier CM, Menard WE. The influence of list format and category headers on age differences in understanding medication instructions. Exp Aging Res. 1998 Jul-Sep;24(3):231-56. doi: 10.1080/036107398244238. PMID 9642551
- [Background] Morrow DG, Leirer VO, Andrassy JM, Tanke ED, Stine-Morrow EA. Medication instruction design: younger and older adult schemas for taking medication. Hum Factors. 1996 Dec;38(4):556-73. doi: 10.1518/001872096778827305. PMID 8976621
- [Background] Morrow D, Leirer V, Sheikh J. Adherence and medication instructions. Review and recommendations. J Am Geriatr Soc. 1988 Dec;36(12):1147-60. doi: 10.1111/j.1532-5415.1988.tb04405.x. PMID 3057053
- [Background] Morrow D, Raquel L, Schriver A, Redenbo S, Rozovski D, Weiss G. External support for collaborative problem solving in a simulated provider/patient medication scheduling task. J Exp Psychol Appl. 2008 Sep;14(3):288-97. doi: 10.1037/a0012809. PMID 18808282
- [Background] Morrow DG, Rogers WA. Environmental support: an integrative framework. Hum Factors. 2008 Aug;50(4):589-613. doi: 10.1518/001872008X312251. PMID 18767520
- [Background] Morrow DG, Weiner M, Young J, Steinley D, Deer M, Murray MD. Improving medication knowledge among older adults with heart failure: a patient-centered approach to instruction design. Gerontologist. 2005 Aug;45(4):545-52. doi: 10.1093/geront/45.4.545. PMID 16051918
- [Background] Morrow DG, Weiner M, Steinley D, Young J, Murray MD. Patients' health literacy and experience with instructions: influence preferences for heart failure medication instructions. J Aging Health. 2007 Aug;19(4):575-93. doi: 10.1177/0898264307304448. PMID 17682075
- [Background] Murray MD, Morrow DG, Weiner M, Clark DO, Tu W, Deer MM, Brater DC, Weinberger M. A conceptual framework to study medication adherence in older adults. Am J Geriatr Pharmacother. 2004 Mar;2(1):36-43. doi: 10.1016/s1543-5946(04)90005-0. PMID 15555477
- [Background] Murray MD, Young J, Hoke S, Tu W, Weiner M, Morrow D, Stroupe KT, Wu J, Clark D, Smith F, Gradus-Pizlo I, Weinberger M, Brater DC. Pharmacist intervention to improve medication adherence in heart failure: a randomized trial. Ann Intern Med. 2007 May 15;146(10):714-25. doi: 10.7326/0003-4819-146-10-200705150-00005. PMID 17502632
- [Background] Paasche-Orlow MK, Parker RM, Gazmararian JA, Nielsen-Bohlman LT, Rudd RR. The prevalence of limited health literacy. J Gen Intern Med. 2005 Feb;20(2):175-84. doi: 10.1111/j.1525-1497.2005.40245.x. PMID 15836552
- [Background] Paasche-Orlow MK, Schillinger D, Greene SM, Wagner EH. How health care systems can begin to address the challenge of limited literacy. J Gen Intern Med. 2006 Aug;21(8):884-7. doi: 10.1111/j.1525-1497.2006.00544.x. No abstract available. PMID 16881952
- [Background] Parker RM, Wolf MS, Kirsch I. Preparing for an epidemic of limited health literacy: weathering the perfect storm. J Gen Intern Med. 2008 Aug;23(8):1273-6. doi: 10.1007/s11606-008-0621-1. Epub 2008 May 2. PMID 18452047
- [Background] Schillinger D, Grumbach K, Piette J, Wang F, Osmond D, Daher C, Palacios J, Sullivan GD, Bindman AB. Association of health literacy with diabetes outcomes. JAMA. 2002 Jul 24-31;288(4):475-82. doi: 10.1001/jama.288.4.475. PMID 12132978
- [Background] Schillinger D, Piette J, Grumbach K, Wang F, Wilson C, Daher C, Leong-Grotz K, Castro C, Bindman AB. Closing the loop: physician communication with diabetic patients who have low health literacy. Arch Intern Med. 2003 Jan 13;163(1):83-90. doi: 10.1001/archinte.163.1.83. PMID 12523921
- [Background] Schillinger D, Wang F, Rodriguez M, Bindman A, Machtinger EL. The importance of establishing regimen concordance in preventing medication errors in anticoagulant care. J Health Commun. 2006 Sep;11(6):555-67. doi: 10.1080/10810730600829874. PMID 16950728
- [Background] Tarn DM, Heritage J, Paterniti DA, Hays RD, Kravitz RL, Wenger NS. Physician communication when prescribing new medications. Arch Intern Med. 2006 Sep 25;166(17):1855-62. doi: 10.1001/archinte.166.17.1855. PMID 17000942
- [Background] Communicating with patients who have limited literacy skills. Report of the National Work Group on Literacy and Health. J Fam Pract. 1998 Feb;46(2):168-76. PMID 9487325
- [Background] Wolf MS, Davis TC, Tilson HH, Bass PF 3rd, Parker RM. Misunderstanding of prescription drug warning labels among patients with low literacy. Am J Health Syst Pharm. 2006 Jun 1;63(11):1048-55. doi: 10.2146/ajhp050469. PMID 16709891
- [Background] Wolf MS, Davis TC, Cross JT, Marin E, Green K, Bennett CL. Health literacy and patient knowledge in a Southern US HIV clinic. Int J STD AIDS. 2004 Nov;15(11):747-52. doi: 10.1258/0956462042395131. PMID 15537462
- [Background] Wolf MS, Davis TC, Osborn CY, Skripkauskas S, Bennett CL, Makoul G. Literacy, self-efficacy, and HIV medication adherence. Patient Educ Couns. 2007 Feb;65(2):253-60. doi: 10.1016/j.pec.2006.08.006. Epub 2006 Nov 21. PMID 17118617
- [Background] Wolf MS, Davis TC, Shrank WH, Neuberger M, Parker RM. A critical review of FDA-approved Medication Guides. Patient Educ Couns. 2006 Sep;62(3):316-22. doi: 10.1016/j.pec.2006.06.010. Epub 2006 Aug 1. PMID 16884888
- [Background] Wolf MS, Davis TC, Shrank W, Rapp DN, Bass PF, Connor UM, Clayman M, Parker RM. To err is human: patient misinterpretations of prescription drug label instructions. Patient Educ Couns. 2007 Aug;67(3):293-300. doi: 10.1016/j.pec.2007.03.024. Epub 2007 Jun 22. PMID 17587533
- [Derived] Chin J, Wang H, Awwad AW, Graumlich JF, Wolf MS, Morrow DG. Health Literacy, Processing Capacity, Illness Knowledge, and Actionable Memory for Medication Taking in Type 2 Diabetes: Cross-Sectional Analysis. J Gen Intern Med. 2021 Jul;36(7):1921-1927. doi: 10.1007/s11606-020-06472-z. Epub 2021 Jan 28. PMID 33507479
- [Derived] Graumlich JF, Wang H, Madison A, Wolf MS, Kaiser D, Dahal K, Morrow DG. Effects of a Patient-Provider, Collaborative, Medication-Planning Tool: A Randomized, Controlled Trial. J Diabetes Res. 2016;2016:2129838. doi: 10.1155/2016/2129838. Epub 2016 Sep 6. PMID 27699179
- [Derived] Morrow DG, Conner-Garcia T, Graumlich JF, Wolf MS, McKeever S, Madison A, Davis K, Wilson EA, Liao V, Chin CL, Kaiser D. An EMR-based tool to support collaborative planning for medication use among adults with diabetes: design of a multi-site randomized control trial. Contemp Clin Trials. 2012 Sep;33(5):1023-32. doi: 10.1016/j.cct.2012.05.010. Epub 2012 Jun 1. PMID 22664648